CLINICAL TRIAL: NCT06649968
Title: Clinical Validation of an Instrumented Glove for Sensorimotor Rehabilitation After Stroke (DESC-Glove)
Brief Title: Clinical Validation of an Instrumented Glove for Sensorimotor Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Cipriani (Other)
Responsible Party: Sponsor-Investigator, Christian Cipriani, Scientific Director, Scuola Superiore Sant'Anna di Pisa
Organization: Scuola Superiore Sant'Anna di Pisa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DESC-Glove Validation; PNC0000007 (Other Grant/Funding Number: Italian Ministry of Research)
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Hand rehabilitation using the device
  Interventions: Device: DESC-Glove (active)
- Sham Group (Sham Comparator): Hand rehabilitation while wearing the device, without providing vibrations to the patients.
  Interventions: Device: DESC-Glove (sham)
- Control Group (Active Comparator): Hand rehabilitation without using the device
  Interventions: Other: Traditional rehabilitation

INTERVENTIONS:
Device: DESC-Glove (active) — Rehabilitation treatment for the upper limb using the DESC-Glove device. The protocol includes 8 exercises, each lasting 2 to 3 minutes. The treatment is conducted daily under the supervision of a therapist and consists of two 20-minute sessions per day, with a 10-minute break in between for neuro-muscular and attentional recovery. The treatment is performed three times a week, totaling 24 sessions over a 4-week period. During each session, patients will wear the DESC-Glove on the affected hand, receiving vibratory stimuli that are synchronized with the exercises being performed.
  Arms: Experimental Group
Device: DESC-Glove (sham) — Rehabilitation treatment for the upper limb using the DESC-Glove device. The protocol includes 8 exercises, each lasting 2 to 3 minutes. The treatment is conducted daily under the supervision of a therapist and consists of two 20-minute sessions per day, with a 10-minute break in between for neuro-muscular and attentional recovery. The treatment is performed three times a week, totaling 24 sessions over a 4-week period. During each session, patients will wear the DESC-Glove on the affected hand, but will not receive any vibratory stimuli.
  Arms: Sham Group
Other: Traditional rehabilitation — Traditional rehabilitation treatment for the upper limb. The protocol includes 8 exercises, each lasting 2 to 3 minutes. The treatment is conducted daily under the supervision of a therapist and consists of two 20- minute sessions per day, with a 10-minute break in between for neuro-muscular and attentional recovery. The treatment is performed three times a week, totaling 24 sessions over a 4-week period. The DESC- Glove will not be used during this treatment.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to evaluate the DESC-Glove, an instrumented glove developed for sensorimotor rehabilitation in individuals recovering from a stroke, utilizing non-invasive vibrational feedback. The primary objective is to assess the technical functionality, safety, and reliability of the device during post-stroke rehabilitation, providing insights for future technical and functional improvements.

The secondary objectives are:

1. To evaluate the usability and acceptability of the device in clinical rehabilitation from the perspectives of both patients and healthcare professionals;
2. To assess the short-term effects of the DESC-Glove on sensorimotor performance and manual dexterity in post-stroke individuals.

To meet the second objective, researchers will compare three groups:

an experimental treatment group (using the DESC-Glove during hand rehabilitation), a sham control group (using the DESC-Glove without vibration), and a conventional control group (receiving hand rehabilitation without the device).

DETAILED DESCRIPTION:
The study is divided into two phases:

Phase 1: Preliminary Investigation of Device Functionality. This phase involves testing the DESC-Glove on 5 patients to assess its initial functionality. Each patient will complete four treatment sessions using the device, focusing on both fine motor exercises for the hand and gross motor exercises for the upper limb. This phase will also help evaluate patient compliance with the rehabilitation treatment on a smaller scale, allowing for a better understanding of the recovery process's duration. During the treatment, patients will wear the DESC-Glove on the affected hand, receiving vibratory stimuli synchronized with the exercises, following the device's operational guidelines.

Phase 2: Multicenter Randomized Controlled Trial (RCT).

In this phase, 42 participants will be recruited and randomly assigned to one of three parallel groups (1:1:1):

The experimental treatment group (using the DESC-Glove), The sham control group (using the DESC-Glove without vibration), and The conventional control group (not using the DESC-Glove). The sample size of 42 (14 participants per group) was chosen following Julious et al. [doi: 10.1002/pst.185], which recommends a minimum of 12 subjects per group for pilot studies. This number was increased to 42 to account for potential dropouts, ensuring robust data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or hemorrhagic stroke confirmed by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI);
* Time from the acute event between 1 and 6 months;
* Mild to moderate impairment of the upper limb, assessed using the Motricity Index (item score for "pinch grip" ≥ 19 and scores for "elbow flexion" and "shoulder abduction" ≥ 14).

Exclusion Criteria:

* Severe behavioral and cognitive disorders (Montreal Cognitive Assessment (MoCA) ≤ 15 ) and/or decreased compliance;
* Spasticity or hypertonia (Modified Ashworth Scale (MAS) > 3) in the affected limb;
* Concurrent participation in a rehabilitation trial that includes treatment training for the upper limb following a stroke;
* Refusal to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Device malfunctioning: number and types of device malfunctions | For both the first and second phase of the study: within one day after each rehabilitation session.
  This outcome measure is designed to systematically document and analyze any malfunctions of the DESC-Glove device throughout the study. All malfunctions will be recorded in detail, including the frequency and type of malfunction. Each issue will be categorized based on the nature of the malfunction, such as hardware failures (e.g., sensor or vibration issues), software, or connectivity problems. This data will be used to assess the overall reliability and functionality of the device, guiding future improvements and treatment efficacy.
Device malfunctioning: number of dropouts device-related | For both the first and second phase of the study: within one day after each rehabilitation session.
  This outcome measure aims to document the number of participants who withdraw from the study specifically due to issues related to the device.

SECONDARY OUTCOMES:
Clinical outcome: Box and Blocks test | For both the first and second phase of the study: baseline assessment (within 3 days before the first rehabilitation session) and final assessment (within 3 days after the last rehabilitation session).
  The Box and Blocks Test is a clinical assessment used to measure manual dexterity and upper limb function. During the test, participants transfer as many small blocks as possible from one compartment of a box to another within 60 seconds. The score is based on the number of blocks successfully moved, reflecting hand coordination and fine motor skills. The test is conducted under three conditions: (a) with the DESC-Glove providing vibratory feedback, (b) with the DESC-Glove not providing vibrations, and (c) without the DESC-Glove altogether
Clinical outcome: Frenchay Arm Test | For both the first and second phase of the study: baseline assessment (within 3 days before the first rehabilitation session) and final assessment (within 3 days after the last rehabilitation session).
  The Frenchay Arm Test (FAT) is an assessment tool designed to measure upper extremity proximal motor control and dexterity during activities of daily living (ADL) in patients with neurological impairments. It focuses on evaluating activity limitations specific to the upper extremities. Each of the test's five items is scored as either a pass (1) or fail (0), with total scores ranging from 0 to 5.
Clinical outcome: Thumb Localizing Test | For both the first and second phase of the study: baseline assessment (within 3 days before the first rehabilitation session) and final assessment (within 3 days after the last rehabilitation session).
  The Thumb Localizing Test is an assessment used to evaluate proprioception and sensory awareness in the hand. During the test, the examiner places the participant's thumb in various positions, either passively or with minimal resistance, while the participant's eyes are closed. The participant is then asked to replicate the position of their thumb with their opposite hand or to indicate the position of their thumb using verbal or tactile cues. It ranges from 0 (normal) to 3 (severely impaired).
Clinical outcome: 5-level EQ-5D | For both the first and second phase of the study: baseline assessment (within 3 days before the first rehabilitation session) and final assessment (within 3 days after the last rehabilitation session).
  The 5-level EQ-5D is a standardized instrument used to measure health-related quality of life. It consists of a descriptive system and a visual analogue scale (VAS). The descriptive system evaluates five dimensions of health - mobility, self-care, usual activities, pain/discomfort and anxiety/depression - each with five levels of severity. The result is calculated by assigning a numerical value to each response level and summing these values across the five items.
Instrumental Outcome: Pick and Lift test | For both the first and second phase of the study: Baseline (within 3 days before the first rehabilitation session); Weekly assessment (within 3 days after the last rehab session of each week).
  The Pick and Lift Test (PLT) assesses the ability of participants to lift a sensorized object using a bi-digit grip with their thumb and index finger. During the test, participants repeatedly lift the object while the levels of force applied during the manipulation tasks are recorded. The PLT is conducted under three conditions: (a) with the DESC-Glove providing vibratory feedback, (b) with the DESC-Glove not providing vibrations, and (c) without the DESC-Glove altogether. This design allows for an evaluation of the impact of vibratory feedback on force application and manipulation skills.
  Such a system is not intended as a clinical validation tool but rather as a means of data acquisition to extract metrics considered standard in the scientific literature regarding motor coordination in manipulation.
Instrumental Outcome: Pick and Place test | For both the first and second phase of the study: baseline assessment (within 3 days before the first rehabilitation session) and final assessment (within 3 days after the last rehabilitation session).
  The Pick and Place Test (PPT) with a fragile object involves performing a series of movements to transfer a fragile item from one side of a barrier to the other. This object walls collapse when the gripping force applied to these walls exceeds a certain threshold. It measures the participant's ability to regulate grip strength and dexterity.
  Such a system is not intended as a clinical validation tool but rather as a means of data acquisition to extract metrics considered standard in the scientific literature regarding motor coordination in manipulation.
Questionnaire: System Usability Scale | For both the first and second phase of the study: final assessment (within 3 days after the last rehabilitation session).
  The system usability scale (SUS) is a simple, ten-item attitude Likert scale giving a global view of subjective assessments of usability. A SUS score can range from 0 to 100, with higher scores indicating better usability. This questionnaire will be evaluated exclusively within the experimental group.
Questionnaire: Gradibility of the Device | For both the first and second phase of the study: final assessment (within 3 days after the last rehabilitation session).
  The Gradibility Questionnaire has been specifically designed to provide a thorough assessment of user experiences. It consists of 13 items that evaluate the usability, acceptability, and satisfaction of users testing the device. This questionnaire will be evaluated exclusively within the experimental group.
Questionnaire: Technology Acceptance Model | For both the first and second phase of the study: final assessment (within 3 days after the last rehabilitation session).
  The Technology Acceptance Model is designed to identify the determinants influencing the acceptance of Robotic and Allied Technology. It comprises four sections: perceived usefulness, ease of use, compatibility, and intention to use. Each question utilizes a 7-point Likert scale, ranging from 1 (worst) to 7 (best). The scoring for each section is calculated as the average of the responses, with scores ranging from 1 (worst) to 7 (best). This questionnaire will be evaluated exclusively within the experimental group.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Fondazione Don Carlo Gnocchi, Polo Specialistico Riabilitativo, Acerenza
  - Fondazione Don Carlo Gnocchi, IRCCS Santa Maria Nascente, Milan
  - Fondazione Don Carlo Gnocchi, Centro Santa Maria della Provvidenza, Roma
  - Fondazione Don Carlo Gnocchi, Centro Santa Maria al Mare, Salerno
  - Fondazione Don Carlo Gnocchi, Polo Specialistico Riabilitativo, Sant'Angelo dei Lombardi
  - Fondazione Don Carlo Gnocchi, Polo Specialistico Riabilitativo, Tricarico

IPD SHARING:
Plan to Share IPD: No